CLINICAL TRIAL: NCT05042765
Title: Entheogen Resurgence - Surveying Entheogen Retreat Participants in Naturalistic Settings
Brief Title: Entheogen Resurgence
Acronym: SERPNTS
Status: Completed | Type: Observational
Sponsor: Vireo Health (Other)
Responsible Party: Sponsor
Other Study IDs: #2021-61137
Record Dates: First submitted 2021-08-30; First posted 2021-09-13 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Psychedelic Experiences
Keywords: Entheogen; Psychedelic; Hallucinogen; Kambo; Ayahuasca; Hapé; Bufo; Sananga

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: self-reported entheogen use — self-reported participation in therapy or a retreat in a naturalistic setting that incorporated the use of entheogens in the past five (5) years

SUMMARY:
For the purpose of this anonymous, observational pilot survey, the investigators will define "entheogens" as substances, generally derived from plants, that are ingested in order to impact one's consciousness for therapeutic, religious, or spiritual purposes. This survey will focus on the naturalistic use of entheogens and other substances including kambo, ayahuasca, hapé, bufo, and sananga typically used in specific cultural and spiritual contexts for healing. There are substantial limitations to what the healthcare community knows about the intentions, motivations, experiences, health behaviors, and demographics of people who decide to participate in entheogen therapy centers or retreats and their willingness to participate in future research studies.

The primary goal of this observational pilot survey is to collect self-reported, anonymous data from people who have opted to participate in entheogen therapy centers and retreats during the last five (5) years on the topics of their initial intentions, motivations, experiences, demographics, and willingness to participate in future entheogen research.

With the support of established therapy and retreat centers, the research team will aim to collect 100 survey responses from unique, unidentified individuals who have participated in some form of entheogen therapy or treatment during the last five (5) years. Those who choose to fill out the survey will be at least 18 years of age, fluent in English, and self-reporting participation in therapy or a retreat which utilized entheogens in a naturalistic setting in the past five (5) years.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Fluent in English
* Self-reported participation in therapy or a retreat in a naturalistic setting that incorporated the use of entheogens in the past five (5) years

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete the online questionnaire
* No self-reported participation in therapy or a retreat in a naturalistic setting that incorporated the use of entheogens in the past five (5) years
* Self-reported participation in therapy or a retreat in naturalistic setting that incorporated the use of entheogens greater than five (5) years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People over the age of 18 years old who are fluent in English and have self-reported participation in entheogen therapy centers or retreats in naturalistic settings during the past five (5) years.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Entheogen Use in Naturalistic Retreat & Therapeutic Settings | Entheogen use will have occured within the last 5 years
  The primary outcome will be self-reported experiences related to entheogen use in naturalistic retreat and therapeutic settings.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Dahmer, ND, Principal Investigator — Resurgent Biosciences, Inc.
Locations (1):
- Vireo Health of New York, Queens, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided